CLINICAL TRIAL: NCT01661153
Title: A Non-interventional Study of Avastin in Combination With Paclitaxel for First Line Treatment in HER2 Negative Metastatic Breast Cancer
Brief Title: An Observational Study of Avastin (Bevacizumab) in Combination With Paclitaxel in First-Line Treatment in Patients With HER2-Negative Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25312
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This prospective observational study will evaluate the use in clinical practice, efficacy and safety of Avastin (bevacizumab) in combination with paclitaxel in first line in patients with HER2-negative metastatic breast cancer. Data will be collected from eligible patients for up to 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Locally recurrent or metastatic breast cancer
* No prior treatment for metastatic or locally recurrent disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2

Exclusion Criteria:

* History or clinical evidence of brain metastases
* Pregnancy
* Uncontrolled hypertension ( systolic > 150 mmHg and/or diastolic > 100 mmHg) or clinically significant (i.e. active) cardiovascular disease
* Major surgical procedure or significant traumatic injury within 28 days prior to enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2-negative breast cancer patients in first-line treatment of metastatic disease
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2011-03-02 (Actual); Primary Completion 2016-09-14 (Actual); Study Completion 2016-09-14 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | approximately 2.5 years

SECONDARY OUTCOMES:
Dosage/schedule/number of cycles of Avastin treatment in clinical practice | approximately 2.5 years
Safety: Incidence of adverse events | approximately 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Croatia (2):
  - Uni Hospital Split; Oncology & Radiotherapy, Split
  - General Hospital Varazdin, Varaždin